CLINICAL TRIAL: NCT01933529
Title: Effects of ARA 290, a Non-hematopoietic Erythropoietin Analogue, on Glucose Tolerance, Insulin Secretion, Insulin Sensitivity and Long-term Glucose Control in Individuals With Prediabetes and/or Drug-naive Type 2 Diabetes; a Phase II Study.
Brief Title: ARA290 in T2D (Effects of ARA 290, an Erythropoietin Analogue) in Prediabetes and Type 2 Diabetes)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Claes-Göran Östenson (Other)
Collaborators: Araim Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Claes-Göran Östenson, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APCP-115; 2012-003207-35 (EudraCT Number)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Type 2; Impaired Glucose Tolerance; Impaired Fasting Glucose
Keywords: diabetes; glucose tolerance; insulin secretion; insulin sensitivity; erythropoietin; inflammation; cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Diabetes Mellitus; Insulin Resistance; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARA 290 (Experimental): ARA 290, 4.0 mg, injected subcutaneously once every morning during 28 days.
  Interventions: Drug: ARA 290
- Placebo (Placebo Comparator): Placebo, injected subcutaneously once every morning during 28 days,
  Interventions: Drug: ARA 290

INTERVENTIONS:
Drug: ARA 290 — ARA 290 is injected s.c. once daily during the study period

SUMMARY:
The purpose of this study is to determine whether a non-hematopoietic erythropoietin analogue, ARA 290, exerts beneficial effects on blood glucose levels and insulin secretion in persons with prediabetes (impaired glucose tolerance, IGT, or impaired fasting glucose, IFG), or drug-naive type 2 diabetes.

The study will also evaluate effects of ARA 290 on insulin sensitivity and serum levels of inflammatory agents, e.g. cytokines. In addition, safety will be monitored by following parameters related to hematology, kidney and liver function and lipid levels.

DETAILED DESCRIPTION:
Aims of the study:

The primary purpose of this double blind study is to determine in individuals with pre-diabetes (IGT, impaired glucose tolerance; or IFG, impaired fasting glucose) and drug-naïve type 2 diabetes whether ARA 290 reduces disease activity by improving oral glucose tolerance, and insulin secretion, and thereby improves long-term glucose control.

Secondary objectives are to evaluate the effects of ARA 290 on insulin sensitivity; serum levels of inflammatory agents, e.g. cytokine levels; serum levels of gluco-regulatory hormones, such as glucagon-like peptide-1 (GLP-1), glucagon; and safety by registering reported adverse events, and by monitoring clinical chemistry parameters related to hematology, kidney function, liver function and lipid levels.

Study Design:

This is a single-center, randomized, double-blind, placebo-controlled clinical trial to evaluate the effects of ARA 290 on glucose homeostasis in persons with pre-diabetes or early, dietary treated type 2 diabetes. The trial has two parallel arms with 12 subjects in each group, and with a 4-week-intervention period. At screening, a baseline investigation will include a physical examination and the following tests: oral glucose tolerance test (OGTT), and glycosylated hemoglobin (HbA1c).

The investigational medicinal product (ARA 290, 4.0 mg) or placebo will be self-administered by a once daily injection s.c. for 28 days. Participating subjects meeting inclusion criteria, and not fulfilling any exclusion criterion on screening, will be randomized double-blind within one week following screening 1:1 to either treatment with ARA 290 or with placebo. Before the first treatment, serum for determination of cytokines, adipokines, and hormones will be collected. Participants will be investigated further with OGTT, HbA1c and clinical assessment after 2 weeks and at study end, after 4 weeks. They should also perform a self-monitoring blood glucose (SMBG) curve once weekly during the treatment period, e.g., altogether 6 blood glucose tests during one day. Four weeks after the last dose, patients will return for HbA1c and fasting blood glucose levels.

The primary endpoint of the study is to test whether there is a significant difference between persons receiving ARA 290 vs. persons receiving placebo in: glucose tolerance, evaluated by OGTT at baseline, and after 2 and 4 weeks. . The secondary endpoints of the study include effects of ARA 290 on: insulin sensitivity, evaluated by HOMA-IR (homeostasis model assessment of insulin resistance); insulin secretion, examined both by measuring the early insulin response (at 15 and 30 min) in OGTT, and using the HOMA-beta (homeostasis model assessment of beta cell function); and long-term glucose control, determined as glycosylated hemoglobin, HbA1c; assessment of serum levels of inflammatory agents, e.g. cytokine levels; serum levels of gluco-regulatory hormones, such as glucagon-like peptide-1 (GLP-1), and glucagon; and safety by registering reported adverse events, and by monitoring clinical chemistry parameters related to hematology, kidney function, liver function and lipid levels.

Patients:

24 patients will be enrolled in one single center; 12 patients will be administered ARA 290 active ingredient product as daily doses for 28 days, and 12 patients will be administered a placebo as daily doses for 28 days. Individuals with IGT (impaired glucose tolerance), IFG (impaired fasting glucose) or drug-naïve type 2 diabetes will be included in the study. The population will consist of individuals of either gender, males aged 40-75 years; women aged 50-75 years and menopausal.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained prior to any trial-related activities
* Meeting criteria for impaired fasting glucose (IFG), impaired glucose tolerance (IGT), IGF+IFG, or type 2 diabetes at the screening OGTT.

IFG = fasting P-glucose 5.6-6.9 mmol/L and 2 hr P-glucose < 7.8 mmol/L; IGT = fasting P-glucose <5.6 mmol/L and 2 hr P-glucose in OGTT 7.8-11.0 mmol/L;diabetes = fasting P-glucose ≥ 7.0 mmol/L and/or 2 hr P-glucose ≥ 11.1 mmol/L.

* Fasting P-glucose ≤ 9 mmol/L.
* BMI (body mass index) ≤ 35 kg/m2.
* Males aged 40-75 years; women aged 50-75 years and in menopause.
* Able to read and understand the written consent form, complete study-related procedures, and communicate with the study staff
* Refrigerator at home for storage of study medication

Exclusion Criteria:

* Anticipated change in concomitant medication that may interfere with blood glucose homeostasis, such as systemic glucocorticoids, non-selective beta blockers and anabolic steroids.
* Anti-diabetic (anti-hyperglycemic) medication of any kind.
* Impaired renal function, defined as S-creatinine ≥ 125 μmol/L for men and ≥ 115 μmol/L for women.
* Impaired hepatic function defined as plasma alanine aminotransferase (P-ALT) ≥ three times the upper reference limit.
* Cardiac disease defined as unstable angina pectoris, or myocardial infarction within the last 6 months, or congestive heart failure NYHA (New York Heart Association) class III or IV.
* Cerebral stroke within the last 6 months.
* Uncontrolled treated or untreated hypertension (systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg).
* Cancer diagnosed and/or treated within the last 5 years.
* Females of childbearing potential.
* Known or suspected abuse of alcohol or narcotic drugs.
* Patients should not have received a vaccination or immunization within the month prior to screening
* The use of Anti-TNF (anti-tumour necrosis factor) therapy or other biological anti-inflammatory agents administered within 3 months prior to screening is not allowed
* The use of erythropoiesis stimulating agents within the two months prior to screening or during the trial is not allowed.
* Administration of an investigational drug trial in the 3 months prior to administration of the initial dose of investigational medicinal product or more than 4 times per year.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
oral glucose tolerance | 28 days
  Oral glucose tolerance tests are performed before and after 2 and 4 weeks of treatment.
  In addition, glucose tolerance will be monitored by checking glycosylated hemoglobin (HbA1c) at the same timepoints, and the participants will perform home blood glucose testing one day every week at home.
Insulin secretion | 28 days
  Plasma insulin levels will be measured at the oral glucose tolerance tests. In addition, insulin secretion will be assessed by HOMA-beta, using fasting glucose and insulin values.

SECONDARY OUTCOMES:
Insulin sensitivity | 28 days
  Insulin sensitivity will be assessed by the HOMA-IR, using fasting glucose and insulin levels at the oral glucose tolerance tests.
Inflammation | 28 days
  Assessment of cytokine levels in serum is reduced by ARA290 treatment.

OTHER OUTCOMES:
Clinical chemistry parameter | 28 days
  Determination of parameters related to hematology, kidney and liver function as well as lipids at baseline and after 28 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Claes-Göran Ostenson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Dept of Endocrinology and Diabetes, Karolinska University Hospital, Stockholm, Sweden